CLINICAL TRIAL: NCT07359365
Title: The Effect of Breathing Exercises on Compassion Fatigue and Work Stress Among Emergency Department Nurses: A Randomized Controlled Trial
Brief Title: The Effect of Breathing Exercises on Compassion Fatigue and Work Tress Among Emergency Department Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Betül Akgün Erol, Master's Student, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CanakkaleOMU-SBF-BAE-01
Record Dates: First submitted 2025-12-21; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Work Stress
Keywords: compassion fatigue
MeSH Terms: conditions — Occupational Stress; Compassion Fatigue | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: This randomized,controlled ,parallel-group study investigates the effects of a breathing exercise on compassion fatiuge and work stress in emergency nurses. Participants are randomly assignefd to an intervention or control group,and outcomes are measured using validated scales
Masking Description: No masking is used in this study. Both participants and researchers are aware of group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing exercise group (Experimental): 32 nurses randomly assigned to the experimental group will receive breathing exercise training. Pre-test and post-test will be conducted to measure compassion fatigue and job stress.
  Interventions: Behavioral: Breathing Exercise Training
- control group (Other): 32 nurses randomly assigned to the control group will not receive breathing exercise training. Pre-test and post-test will be conducted to measure compassion fatigue and job stress.
  Interventions: Other: usual care

INTERVENTIONS:
Behavioral: Breathing Exercise Training — Participants in the experimental group will receive training on proper breathing techniques and breathing exercise methods. Each session will last 30-40 minutes. Sessions will be conducted twice a week for a total of 4 weeks.
  Arms: Breathing exercise group
Other: usual care — No intervention will be applied. Participants in the control group will continue their usual routine.
  Arms: control group

SUMMARY:
The purpose of this randomized controlled study is to examine the effect of breathing exercises on compassion fatigue and work stress among emergency department nurses

DETAILED DESCRIPTION:
"This study will be conducted with nurses working in the emergency department. Participants will be randomly assigned to either an intervention group receiving breathing exercise training or a control group. Data will be collected using a sociodemographic data form and validated scales measuring work stress and compassion fatigue. The aim of the study is to evaluate the effect of breathing exercises on work stress and compassion fatigue levels among emergency department nurses."

ELIGIBILITY:
Inclusion Criteria:

* Currently employed as an emergency department nurse.
* No diagnosed psychiatric disorders.
* No prior participation in breathing exercise programs.

Exclusion Criteria:

* Presence of respiratory system disease.
* Physical conditions that prevent participation in breathing exercises.
* Working outside the emergency department.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Compassion Fatigue Score (Adams ve ark,2006) | Baseline and 4 weeks after ınvertıon
  The level of compassion fatigue among emergency department nurses will be assessed using the Compassion Fatigue Scale (Figley, 2006). This is a Likert-type scale ranging from 1 ("Never") to 10 ("Very Often"). The scale consists of two subdimensions: secondary traumatic stress and occupational burnout. Specifically, items C, E, H, K, and L assess secondary traumatic stress, while items A, B, D, F, G, I, K, and M assess occupational burnout.
  The internal consistency of the subdimensions, measured by Cronbach's alpha, ranges from 0.80 to 0.90, indicating sufficient reliability. Total scores on the scale range from 13 to 130, with higher scores reflecting higher levels of compassion fatigue experienced by the individual. Measurements will be taken at baseline and at 8 weeks after the intervention.
Work Stress Score (Nurse Work Stress Scale, Gray-Toft & Anderson,(1981); validated in Turkey by Mert et al.,(2021( | Baseline and 4 weeks after ınvertıon
  Work-related stress among emergency nurses will be measured with the 34-item Nurse Work Stress Scale (Gray-Toft & Anderson, 1981; validated in Turkey by Mert et al., 2021). The scale has seven subdimensions: uncertainty concerning treatment (items 1-8), workload (items 9-14), patient death (items 15-19), conflict with physicians (items 20-24), conflict with other nurses (items 25-29), inadequate support (items 30-32), and suffering patient (items 33-34). Items are scored on a 4-point Likert scale (1=Never, 2=Sometimes, 3=Often, 4=Very Often). Subdimension reliability ranges from α=0.65 to α=0.89. Total scores are summed; higher scores indicate higher work-related stress.

CONTACTS AND LOCATIONS:
Overall Officials: gülnur A akkaya, Principal Investigator — Çanakkale onsekiz mart universty
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No